CLINICAL TRIAL: NCT06887166
Title: Efficacy of Platelet-rich Plasma on Perianal Wound Healing After Anal Fistulotomy: A Randomized Controlled Clinical Trial
Brief Title: Platelet- Rich Plasma Injection
Acronym: prp
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mansoura University (Other)
Responsible Party: Principal Investigator, Mirna Mohamed Elsaid, assistant lecturer of general surgery, Mansoura University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PRP in perianal wound healing
Record Dates: First submitted 2025-03-14; First posted 2025-03-20 (Actual); Last update posted 2025-03-25 (Actual); Status verified 2025-03

CONDITIONS: Wound Healing; Anal Fistula
Keywords: prp; wound healing; perianal wounds
MeSH Terms: conditions — Rectal Fistula; Insomnia, Fatal Familial

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- platelet rich plasma (Active Comparator): will be injected with PLATELT RICH PLASMA in addition to the usual surgery
  Interventions: Procedure: Platelet Rich Plasma
- control (No Intervention): a control group will be treated with the usual surgery only

INTERVENTIONS:
Procedure: Platelet Rich Plasma — injection of PRP IN PERIANAL WOUNDS AFTER FISTULOTOMY OPERATIONS
  Arms: platelet rich plasma

SUMMARY:
This randomized controlled study aims to investigate the effect of injection of platelet rich plasma on the postoperative outcome of perianal wound after anal fistula surgery in terms of healing time, reduction in wound size, pain score , and therefore quality of patients' life.

DETAILED DESCRIPTION:
Fistula-in-ano is an epithelial-lined tract connecting the anal canal to the perianal skin. Most commonly, it affects people in the third to fifth decades of life.

Anal fistula arise spontaneously, when it is referred to as idiopathic or cryptoglandular, or as a result of an underlying pathology, such as inflammatory bowel disease, malignancy, trauma or irradiation.

The majority of anal fistula often occurs following anorectal abscess. An anorectal abscess occurs when an anal gland becomes obstructed, resulting in infection and abscess formation. One-third of patients undergoing incision and drainage of an anorectal abscess will later develop a fistula. Thirty to 70% of patients diagnosed with an anorectal abscess will already have a fistula present on exam.

According to the relation of fistulous track to the sphincter complex, anal fistulas can be classified as simple or complex. Simple anal fistula includes low transsphincteric and intersphincteric fistulas that cross less than 30% of the external sphincter fibers. On the other hand, complex anal fistulas comprise, high transsphincteric fistulas, suprasphincteric, extrasphincteric fistulas, and horseshoe fistulas.

Patients with anal fistula often complain of perianal cellulitis, anorectal pain, pruritus ani, smelly or bloody drainage of pus, and in some cases difficulty controlling bowel movements.

In the long term, it results in significant morbidity through development of recurrent abscesses due to occlusion of the external opening leading to episodes of fever, exquisite perianal pain and discharge, and financial implications through time off work and repeated hospital admissions.

An anorectal fistula is a clinical diagnosis, but imaging is beneficial in determining the course of a fistulous tract or determining its etiology. Imaging studies include endo-anal ultrasound, CT pelvis, CT-fistulography, and MRI of the pelvis. Still, in general, an exam under anesthesia is typically indicated to identify the fistulous tract using a lacrimal probe and methylene blue or hydrogen peroxide.

The treatment for anal fistulae depends on etiology. While the treatment of simple anal fistula is usually straightforward with fistulotomy being recommended as the first line of treatment; the management of more complex cases requires more sophisticated treatments aiming to preserve the anal sphincters and to eradicate the fistulous track. Surgery for complex anal fistula includes the placement of seton, anal advancement flap, laser ablation, fistula plug, and video-assisted anal fistula treatment.

Postoperative pain and delayed wound healing are the main complications following anal surgery associated with poor quality of life.

Platelet-rich plasma (PRP) is an endogenous therapeutic technology that is gaining interest in regenerative medicine due to its potential to stimulate and accelerate tissue healing. PRP is defined as an autologous biological product derived from the patient's blood, and in which after a centrifugation process a plasma fraction is obtained with a platelet concentration higher than that in circulating blood.

Platelets play a crucial role in the wound healing process thanks to their hemostatic function and presence of cytokines and growth factors.

A recent randomized controlled clinical trial investigated the effect of injection of Platelet-rich plasma in patients with open surgery for pilonidal sinus disease in postoperative recovery. It showed that PRP application improves postoperative recovery in that it speeds patients' return to daily activities, reduces their pain scores and increases their quality of life.

No previous studies were designed to investigate the effect of platelet rich plasma injection on perianal wound healing. Our hypothesis entails that platelet rich plasma decrease the complication rate of anal fistula surgery which includes chronic draining wound and pain therefore accelerate the recovery of the patient, return to work and improve the quality of life.

ELIGIBILITY:
Inclusion Criteria:

1. Both genders
2. Aging between 18-65 years
3. Presented by simple anal fistula (subcutaneous, intersphincteric, or low trans-sphicnteric involving less than 30% of external anal sphincter fibers)

Exclusion criteria:

1. Patients with associated anorectal pathology such as anal fissure, hemorrhoids, rectal prolapse, neoplasm, solitary rectal ulcer, inflammatory bowel diseases.
2. Patients on long-acting corticosteroids or immunosuppressive drugs
3. Patients having connective tissue diseases
4. Patients with complex anal fistula.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2023-07-14 (Actual); Primary Completion 2024-07-14 (Actual); Study Completion 2024-08-05 (Actual)

PRIMARY OUTCOMES:
complete wound healing | from day 1 post operative to maximally 6 months
  duration in days required to achieve complete healing of the anal wound in both groups on postoperative follow-up

SECONDARY OUTCOMES:
pain score | from 6 hours postoperative to 2 months
  pain score assessed using Visual Analogue Scale; it measures pain intensity; where 0 ('no pain') and 10 ('pain as bad as it could possibly be').

CONTACTS AND LOCATIONS:
Overall Officials: emad a proffesor, Study Chair; samy e associate professor, Study Director; ahmed h lecturer, Study Director
Locations (1):
- Mansoura University Hospital, Al Mansurah, Dakahliya, Egypt

IPD SHARING:
Plan to Share IPD: No
data is available with corresponding author on request

REFERENCES:
- [Background] Boztug CY, Karaagac Akyol T, Benlice C, Koc MA, Doganay Erdogan B, Ozcebe OI, Kuzu MA, Akyol C. Platelet-rich plasma treatment improves postoperative recovery in patients with pilonidal sinus disease: a randomized controlled clinical trial. BMC Surg. 2021 Oct 21;21(1):373. doi: 10.1186/s12893-021-01370-5. PMID 34670534
- See also: Platelet-rich plasma treatment improves postoperative recovery in patients with pilonidal sinus disease: a randomized controlled clinical trial — https://bmcsurg.biomedcentral.com/articles/10.1186/s12893-021-01370-5